CLINICAL TRIAL: NCT03474536
Title: Clinical Impact of Concentration and Affinity of HLA-DQ Antibodies in Lung Transplantation - AFFIHLA-P
Brief Title: Quantitative Parameters of HLA-DQ Antibodies in Lung Transplantation
Acronym: AFFIHLA-P
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/35
Record Dates: First submitted 2018-03-05; First posted 2018-03-22 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplantation; Antibody Mediated Rejection; Chronic Lung Allograft Dysfunction
Keywords: Lung transplantation; HLA antibodies; concentration; affinity; surface plasmon resonance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to compare the quantitative parameters of de novo anti-HLA DQ Donor Specific Antibodies (DSA), determined at the time of their discovery by surface plasmon resonance (SPR), between recipients that developed a Chronic Lung Allograft Dysfunction (CLAD) for the 2 years following DSA apparition and those who did not. If concentration, kinetics and/or affinity parameters of anti-DQ DSA are associated with CLAD development, new, non-invasive prognostic biomarkers of humoral rejection in lung transplantation will be discovered .

DETAILED DESCRIPTION:
After lung transplantation the production of de novo DSA directed against HLA-DQ molecules is associated with CLAD and graft loss. The most used assay for serum DSA detection is the Single Antigen Luminex® (SAG), which provides a semi-quantitative fluorescence value, the MFI, used as a surrogate of DSA "strength". But MFI is not perfectly associated with CLAD development. We developed a method using SPR allowing the concentration, kinetics (ka, kd) and affinity parameters (KD) of anti-DQ DSA to be determined. These quantitative parameters could represent biomarkers finely associated with CLAD. The way this parameters evolve (stability, increase or decrease) with time could also impact on DSA pathogenicity. We will compare the quantitative parameters of de novo anti-HLA DQ DSA, determined at the time of their discovery, between recipients that developed a CLAD for the 2 years following DSA apparition, and those who did not. The association between quantitative parameters of DSA and graft loss, their evolution and its association with CLAD and graft loss, and their correlation with SAG MFI will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patient transplanted between 01/01/2001 and 31/07/2016
* Patient with immunodominant anti-HLA DQ de novo DSA developed before 08/2016
* Patient for who sufficient remaining serum quantity is available in usual care biobank
* non-opposition of the patient

Exclusion Criteria:

* preformed DSA at the transplantation;
* Non immunodominant DQ DSA ;
* Insufficient serum quantity in usual care biobank
* Inability to determine the date of DSA apparition at around one year
* opposition of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 122 patients with lung transplantation at University Hospital of Bordeaux and 4 departments of lung transplantation from Paris (Marie Lannelongue, Foch, Bichat and HEGP hospitals
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
CLAD development | 2 years
  CLAD development within the 2 years following DSA apparition

SECONDARY OUTCOMES:
raft loss up to 5 years following DSA apparition | 6 months, 1 year, 2 years, 5 years
  Graft loss up to 5 years following DSA apparition, defined by re-transplantation or recipient's death
CLAD development | 6 months
  CLAD development 6 months following DSA apparition
CLAD development | 1 year
  CLAD development 1 year following DSA apparition

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Bordeaux, Bordeaux
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - Hôpital Européen Georges Pompidou, Paris
  - AP-HP Hôpital Bichat, Paris
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No